CLINICAL TRIAL: NCT04395690
Title: Prospective Randomized Multicenter Study Between Two Anesthetic Techniques for Implant Placement in the Posterior Mandible
Brief Title: Comparing Two Anesthetic Techniques for Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator, Aula Dental Avanzada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADA-1
Record Dates: First submitted 2020-05-12; First posted 2020-05-20 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Edentulous Jaw; Dental Implant; Anesthesia, Local
Keywords: Anesthesia; Inferior Alveolar Block Nerve; Infiltration; Dental implant; Mandible
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: 48 receiving infiltrative anesthesia and 48 patients receiving Inferior Alveolar Block Nerve anesthesia. (n=96)
Who Masked: Participant, Investigator
Masking Description: Patients were not told what type of anesthesia was being used and surgeons obtains the method of anesthesia to be used in this particular patient thirty minutes before intervention started.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferior Alveolar Block Nerve (IABN) (Active Comparator): Inferior Alveolar Block Nerve (IABN) anesthesia technique before posterior mandibular implant placement.
  Interventions: Procedure: Dental Implant Placement in the posterior mandible
- Infiltration (INF) (Experimental): Infiltration (INF) anesthesia technique before posterior mandibular implant placement.
  Interventions: Procedure: Dental Implant Placement in the posterior mandible

INTERVENTIONS:
Procedure: Dental Implant Placement in the posterior mandible — Surgery done in the posterior mandible with missing teeth for placing dental implants.
  Other Names: Implant surgery

SUMMARY:
To evaluate in a comparative way the patient's perception in implant surgery in the posterior mandibular quadrants depending on whether the operation is performed under trunk anaesthesia or infiltrative anaesthesia, in both cases with Articaine.

Randomized and multicenter prospective study to be developed in eight centers with similar socio-professional characteristics, with the same operative protocol.

A significant sample of patients will be randomized to undergo the same intervention (surgery to place implants in the posterior mandible) under one or another type of anesthesia (inferior alveolar block nerve or infiltrative) and data will be collected using a Numerical Rate scale on four occasions (after the incision, after drilling, after suturing and after 12h).

DETAILED DESCRIPTION:
The optimal anesthesia for posterior mandibular implant surgery remains controversial and dependent on operator's preferences. Although not evidence-based, most operators usually avoid infiltration anesthesia in the posterior mandible due to its uncertain efficacy. However, various comparative studies with articaine 4% have not found differences between infiltration (INF) and inferior alveolar nerve block (IANB) but current research is still conflicting.

Infiltration anesthesia is easier for the operator and more tolerable for the patient. Should it were sufficient for surgical procedures in the posterior mandible it could become the first option in routine surgeries.

The purpose of this prospective, randomized and multicenter study is to clarify the efficacy of infiltration anesthesia for placing implants in the posterior mandible.

The study will take place in eight centers with similar socio-professional characteristics and the same operative protocol. The study has been approved by the Ethical Research Committee of the University Hospital of San Juan (Alicante, Spain).

On a significant sample of patients (96n) that meet the in-exclusion criteria, the same intervention (implant placement surgery in posterior area of the mandible) has been carried out randomly (List Randomizer, www.random.org/lists) with one or another type of anesthesia (group A: IANB or group B: INF).

Data of pain perception from patients were collected intraoperatively, by means of a Numerical Rating Scale, in three moments (after incision, after drilling, after suturing) and global satisfaction one week post surgery.

Five confounding variables were also recorded, gender, use of release incision, number of implants placed, wether or not Guided Bone Regeneration (GBR) was applied and the distance from the implant apex to the mandibular canal. A non-parametric statistical analysis was applied.

ELIGIBILITY:
Inclusion Criteria:

* Patient in health status American Society of Anesthesiologists (ASA) I and ASA II
* Any age and gender
* Unitary or multiple posterior mandibular edentulism.
* Need to replace at least one implant and at least 2mm distal to mental foramen
* Absence of orofacial neurological symptoms

Exclusion Criteria:

* Any contraindication for implant surgery.
* Hypersensitivity to any of the products used in the study
* ASA patients ≦ II
* Pharmacological allergies that contraindicate the intervention
* Patients medicated with sedatives or analgesics up to 24h before the intervention
* Psychotropic drug abuse or medication that may alter painful perception 15 days before the intervention
* Pregnant or nursing women
* Interventions with conscious sedation
* Women on contraceptive treatment
* Bisphosphonate-treated patients
* Pathological mental state (dementia, psychosis)
* Severe dental anxiety
* Lack of collaboration
* Signs of infection in the area to be operated
* Unconventional surgical requirements (split crest, vertical regeneration, block graft, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Esteve-Pardo, DDS, Principal Investigator — Aula Dental Avanzada
Locations (8):
- Spain (8):
  - Clinica Dental José Antonio Sánchez Nicolás, Cabezo de Torres, Alicante
  - GMD Ambrosio Bernabeu, Elche, Alicante
  - Salgado Dental Institute, Orihuela, Alicante
  - LG Dental, San Pedro del Pinatar, Murcia
  - Clínica Dental Esteve, Alicante
  - TREES Clinica Dental, Cartagena
  - Clínica Dental García Vega, Madrid
  - Clinica Dental Amigó, Valencia

IPD SHARING:
Plan to Share IPD: No
No plan to share with other researches.

REFERENCES:
- [Background] Kim S, Lee YJ, Lee S, Moon HS, Chung MK. Assessment of pain and anxiety following surgical placement of dental implants. Int J Oral Maxillofac Implants. 2013 Mar-Apr;28(2):531-5. doi: 10.11607/jomi.2713. PMID 23527356
- [Background] Alghamdi AS. Pain sensation and postsurgical complications in posterior mandibular implant placement using ridge mapping, panoramic radiography, and infiltration anesthesia. ISRN Dent. 2013 May 21;2013:134210. doi: 10.1155/2013/134210. Print 2013. PMID 23762571
- [Background] Bataineh AB, Alwarafi MA. Patient's pain perception during mandibular molar extraction with articaine: a comparison study between infiltration and inferior alveolar nerve block. Clin Oral Investig. 2016 Nov;20(8):2241-2250. doi: 10.1007/s00784-016-1712-8. Epub 2016 Jan 21. PMID 26791025
- [Background] Garcia-Blanco M, Gualtieri AF, Puia SA. A randomized controlled trial comparing nerve block and mandibular infiltration techniques in posterior mandible implant surgeries. J Clin Exp Dent. 2018 Oct 1;10(10):e1003-e1010. doi: 10.4317/jced.54330. eCollection 2018 Oct. PMID 30386507
- [Background] Etoz OA, Er N, Demirbas AE. Is supraperiosteal infiltration anesthesia safe enough to prevent inferior alveolar nerve during posterior mandibular implant surgery? Med Oral Patol Oral Cir Bucal. 2011 May 1;16(3):e386-9. doi: 10.4317/medoral.16.e386. PMID 21196835
- [Background] Heller AA, Shankland WE 2nd. Alternative to the inferior alveolar nerve block anesthesia when placing mandibular dental implants posterior to the mental foramen. J Oral Implantol. 2001;27(3):127-33. doi: 10.1563/1548-1336(2001)0272.3.CO;2. PMID 12500871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population was composed by all patients scheduled for the placement of implants in the area distal to the mental foramen, in each of the 8 participating centers, between January 4, 2019 and March 7, 2021.
Pre-assignment Details: Two patients, 1 of each group, out of the initial 96 included in the study, had to be excluded from the analysis classified as "anesthetic failures". In the IANB group, 1 nerve block resulted in being ineffective and the operator had to use an intraosseous technique. In the INF group, 1 patient needed additional injections to continue the surgery and was also excluded.
Period: Overall Study
Arm/Group | Inferior Alveolar Block Nerve (IABN) | Infiltration (INF)
Started | 48 | 48
Completed | 47 | 47
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants were adult patients of any age and gender, in health status ASA I or ASA II, with posterior mandibular edentulism, requiring to replace at least one implant and at least 2 mm distal to mental foramen (in positions 45, 46, 47, 35, 36, 37, according to the FDI notation) and without contraindication for implant surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Inferior Alveolar Block Nerve (IABN) | Infiltration (INF) | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 40 | 79
  >=65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 24 | 17 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 47 | 47 | 94
Pain perception [Median (Inter-Quartile Range); unit: units on a scale] — Patients' perceived pain by a numerical rating scale (NRS).
  units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: Pain Perception by Numerical Rating Scale
Description: Pain perception by the patient during surgical procedure, being 0 no pain at all, 1-3 mild discomfort, 4-7 moderate pain and 7-10 intense pain
Time Frame: Pain perceived by the patient during surgery after the incision, the osteotomy and the suture
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Inferior Alveolar Block Nerve (IABN) | Infiltration (INF)
Number analyzed (Participants) | 47 | 47
score on a scale | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Satisfaction of the Patient by Numerical Rating Scale
Description: Patients satisfaction 12 hours after operation, being 0 not satisfied at all, and 10 very satisfied
Time Frame: Satisfaction of the patient 12 hours after surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inferior Alveolar Block Nerve (IABN) | Infiltration (INF)
Number analyzed (Participants) | 47 | 47
score on a scale | 9 (1) | 8.8 (1.7)

ADVERSE EVENTS:
Time Frame: 7 days
Description: Other (Not Including Serious) such as inferior alveolar nerve injury or local anesthetic toxicity.
Arm/Group | Inferior Alveolar Block Nerve (IABN) | Infiltration (INF)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT04395690/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT04395690/ICF_002.pdf